CLINICAL TRIAL: NCT04768244
Title: Impact of Maternal SARS-CoV-2 Infection and Vaccination on Breast Milk Antibodies, Milk Bioactive Compounds and Maternal-child Health (MilkCORONA)
Brief Title: Impact of Maternal COVID-19 Disease on Breast Milk and Infant Health
Acronym: MilkCorona
Status: Completed | Type: Observational
Sponsor: Institute of Agrochemistry and Food Technology, National Research Council (Other Government)
Collaborators: Hospital Universitario La Fe (Other); Instituto de Investigacion Sanitaria INCLIVA (Other); Hospital Clínico Universitario de Valencia (Other); Hospital Universitario Doctor Peset (Other); Universidad de Granada (Other); Universitat Jaume I (Other); Hospital Sant Joan de Deu (Other); Fetal Medicine Research Center, Spain (Other); Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Principal Investigator, Maria Carmen Collado, PhD, Research Scientist, Institute of Agrochemistry and Food Technology, National Research Council
Other Study IDs: covid1
Record Dates: First submitted 2021-02-10; First posted 2021-02-24 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Covid19
Keywords: Breast milk; Microbiota; Sars-CoV-2; metabolites; immune compounds; infant growth and development
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID19: - Women with SARS-CoV-2 infections
  Interventions: Other: maternal SARS-CoV-2 infection

INTERVENTIONS:
Other: maternal SARS-CoV-2 infection — positive PCR in nasopharinx and/or presence of antibodies in serum

SUMMARY:
prospective multicenter study The main aim is to study the impact of maternal COVID-19 on breast milk immune, microbiological, and metabolic profile and infant growth and development

ELIGIBILITY:
Inclusion Criteria:

* pregnant or nursing women with positive PCR for SARS-CoV-2 in nasopharynge and/or presence of SARS-CoV-2 antibodies in serum determined in hospitals

Exclusion Criteria:

* aggravation of symptomatology requiring specific treatment and/or hospitalization

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women at the end of the pregnancy and also, lactating women
Study Population: Women with SARS-CoV-2 infection at the end of pregnancy, before delivery following hospitals COVID19 screening protocols.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 RNA | 1 month
  levels of viral RNA from SARS-CoV-2 in breast milk

SECONDARY OUTCOMES:
breast milk immune | 1st year
  interleukines, cytokines and growth factors, immunoglobulins
breast milk microbiota | 1st year
  microbiota composition and diversity
breast milk metabolite | 1st year
  metabolite profile
infant microbiota | 1st year
  infant microbiota profile
infant growth and development | 1st year
  z-scores growth curves

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Fundacion Investigacion Sanitaria INCLIVA, Valencia
  - Hospital Universitario y Politecnico la Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bauerl C, Randazzo W, Sanchez G, Selma-Royo M, Garcia Verdevio E, Martinez L, Parra-Llorca A, Lerin C, Fumado V, Crovetto F, Crispi F, Perez-Cano FJ, Rodriguez G, Ruiz-Redondo G, Campoy C, Martinez-Costa C, Collado MC; MilkCORONA study team. SARS-CoV-2 RNA and antibody detection in breast milk from a prospective multicentre study in Spain. Arch Dis Child Fetal Neonatal Ed. 2022 Mar;107(2):216-221. doi: 10.1136/archdischild-2021-322463. Epub 2021 Aug 20. PMID 34417223